CLINICAL TRIAL: NCT06162130
Title: Investigation of Muscular Activations During Eccentric Quadriceps Exercises
Brief Title: Muscular Activations During Eccentric Quadriceps Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Elif AYGUN POLAT, PhD, Ordu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ODUSBFFTR-ELIFAYGUNPOLAT-001
Record Dates: First submitted 2023-12-01; First posted 2023-12-08 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: ACL Injury; Sport Injury; Sports Physical Therapy; Muscle Weakness
Keywords: Electromyography; Exercise Theraphy; Eccentric Exercises; Quadriceps; Muscle Activity
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Other (Experimental): female athletes
  Interventions: Diagnostic Test: Eccentric quadriceps exercises

INTERVENTIONS:
Diagnostic Test: Eccentric quadriceps exercises — The activation of the vastus medialis, vastus lateralis, and rectus femoris muscles will be measured using surface electromyography (sEMG) during four distinct quadriceps eccentric exercises: Reverse Nordic, Pistol squat, Suspension-based Bulgarian split squat, and Bulgarian split squat. Participants will be instructed to perform three successful repetitions for each exercise. A 30-second break will be provided between each repetition, and there will be a minimum of 10 minutes of rest between each of the four exercises. Due to the belief that fatigue could impact exercise performance, the modified Borg scale will be used to ensure that fatigue does not occur before each exercise. Exercise recording will commence when scores reported using the modified Borg scale are 1 or lower.

SUMMARY:
The aim of this study is to investigate muscular activations during various quadriceps exercises commonly used in clinical settings.

DETAILED DESCRIPTION:
The quadriceps muscle is known to be crucial for the dynamic control of the lower extremity, and weakness in this muscle can lead to strategies that may result in injury. Therefore, acquiring optimal quadriceps muscle strength is essential not only for preventing lower extremity injuries but also for enabling individuals to fully return to activities after an injury.

Despite the existence of various eccentric quadriceps exercises in the literature, there is a lack of consensus on their comparative effectiveness. Hence, there is a requirement for research to explore the effectiveness of different eccentric quadriceps exercises. The objective of this study is to compare the muscular activation of the quadriceps muscle during four distinct eccentric quadriceps exercises using surface electromyography (sEMG) devices

ELIGIBILITY:
Inclusion Criteria:

Being a licensed athlete in one's own field, Having been engaged in sports for at least 2 years

Exclusion Criteria:

Individuals with any musculoskeletal injury history in the lower extremities and trunk that could impede exercise within the last year, Individuals with systemic, neurological, and/or cognitive issues, Individuals experiencing pain in the lower extremities and trunk during exercises

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Surface EMG Measurement | in an average of one hour
  During data collection, the EMG Noraxon MiniDTS system (Noraxon Inc.) was used to measure the signals from the muscle. Additionally, the participants were video-recorded to prevent any potential mistakes that might have gone unnoticed during the activities.
Normalization of Surface EMG | in an average of one hour
  To normalize the EMG data obtained during the exercises, MVIC will be performed for each muscle using an isokinetic dynamometer. Participants will be shown a video demonstrating the movement for MVIC, and before the test, they will be asked to warm up for 5 minutes on a treadmill at submaximal speed and then perform the movement. To ensure electromyography (EMG) normalization, participants will be asked to perform 3 repetitions, and the average of these three values will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Elif AYGUN POLAT, PhD, Principal Investigator — Ordu University; Nevin A. GUZEL, Prof, Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.